CLINICAL TRIAL: NCT02640599
Title: The Effect of Vestibular and Exertion Training on Gait, Balance and Dizziness in Individuals With Concussion
Brief Title: Stationary Bike Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-01231
Record Dates: First submitted 2015-12-18; First posted 2015-12-29 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Vertigo; Concussion; Dizziness
Keywords: Vestibular; Rehabilitation
MeSH Terms: conditions — Vertigo; Brain Concussion; Dizziness | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Rehabilitation + Areobic Exercise (Experimental)
  Interventions: Other: Vestibular Rehabilitation + Aerobic Exercise
- Vestibular Rehabilitation (Active Comparator)
  Interventions: Other: Vestibular Rehabilitation

INTERVENTIONS:
Other: Vestibular Rehabilitation + Aerobic Exercise — Subjects in the experimental group will undergo traditional Vestibular Rehabilitation as well as participate in an aerobic exercise training program.
  Arms: Vestibular Rehabilitation + Areobic Exercise
Other: Vestibular Rehabilitation — The control group will receive standard care which includes participation in vestibular physical therapy treatments 1-2 times per week.
  Arms: Vestibular Rehabilitation

SUMMARY:
Investigators will use a stationary bike protocol to investigate whether patients with post concussion syndrome benefit from adding exertion training to a vestibular rehabilitation program.

Investigators examine the effect of aerobic exercise testing and training on individuals with concussion who are currently experiencing symptoms and examine the effect of aerobic exercise in combination with traditional vestibular rehabilitation.

DETAILED DESCRIPTION:
This is a randomized controlled single blind pilot study testing the hypothesis that the combination of aerobic exercise plus vestibular rehabilitation will result in greater reduction of symptoms of dizziness and imbalance compared to vestibular rehabilitation alone.

ELIGIBILITY:
Inclusion Criteria:

1. History of concussion >14 days, <6 months
2. One or more of the following symptoms after most recent head injury: headache, dizziness, fatigue, irritability, insomnia, concentration or memory difficulty)
3. Age range - 18-70
4. Access to stationary bicycle
5. Ability to read and write sixth grade English

Exclusion Criteria:

1. Inability to participate in aerobic exercise for any reason
2. Pre-existing or current neurological or autonomic disease including persistent symptoms form previous concussion
3. Major depressive disorder
4. Litigation
5. Increased cardiac risk
6. Currently taking, Beta Blockers, or Anticonvulsants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-11-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Changes in Visual Analog Scale (VAS) of Dizziness Score | change in VAS of Dizziness Score from initial evaluation to week 6
Changes in Dizziness Handicap Inventory (DHI) Score | change in DHI Score from initial evaluation to week 6
  25-item scale that addresses the functional, emotional, and physical components of dizziness. Higher scores indicate greater handicap (range, 0 - 100)
Change in the number of symptoms on checklist of the Sports Concussion Assessment Tool | change in symptoms from initial evaluation to week 6
Changes in balance Error Scoring System (BESS) score | change in (BESS) Score from initial evaluation to week 6
  requires participants to maintain balance with eyes closed with their hands on their iliac crests under six different surface conditions. Number of errors in each trial are added together to obtain a total score (out of 60).
Changes in Dynamic Visual Acuity (DVA) Score | change in DVA Score from initial evaluation to week 6
  instrumented, objective assessment of vestibulo-ocular reflex (VOR) function in response to head movement. The Dynamic Visual Acuity Test assesses visual acuity during head movement relative to baseline static visual acuity
Changes in Sport Concussion Assessment Tool (SCAT-3) Score | change in (SCAT-3) from initial evaluation to week 6
  22 item postconcussion symptom scale using a seven point Likert rating. This scale provides an assessment of symptoms endorsed, along with a severity score. The maximum symptom score is 22, the symptom severity score is obtained by summing the rated symptom score for each symptom (maximum score 132).
Functional Gait Assessment | change in gait from initial evaluation to week 6
  10-item test that measures gait with a narrow base of support, gait with eyes closed, ambulating backwards, as well as ambulation with head turns. The maximum score is 30. Higher scores indicate better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Denham, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States